CLINICAL TRIAL: NCT05375877
Title: Evaluation of a Digital Care System in the Follow-Up Care of Atrial Fibrillation Patients
Acronym: EDVIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: iATROS GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2022-02-14; First posted 2022-05-17 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Cardiovascular Diseases; Atrial Fibrillation
Keywords: eHealth; cardiology; atrial fibrillation
MeSH Terms: conditions — Cardiovascular Diseases; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, longitudinal study with event-based design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital eHealth platform with connected mobile 1-lead ECGs + Standard of Care (Other): Patients will be fitted with a 1-channel ECG monitor after inclusion in the study and discharged to post ablation care. Here, ECGs are recorded regularly until the occurrence of an arrhythmic event. After the occurrence of an event, a discussion with the investigator will be performed. Interim medical contacts will be limited to the agreed-upon follow-up appointments for the long-term ECGs and other appointments routinely scheduled in the patient's care according to the Standard of Care.
  long-term ECGs at defined time points
  Interventions: Device: iATROS

INTERVENTIONS:
Device: iATROS — The digital eHealth platform of iATROS in combination with a wearable will be used independently by the subjects of the study. In particular, the reminder function is used to remind patients to record their ECGs, take medication and perform other tasks they may have created themselves, or to use other iATROS functions, such as teleconsultation or remote medical data reporting. Furthermore, the designed training program for atrial fibrillation patients teaches them how to deal with their own disease.
  If unhealthy or dangerous vital signs are detected during the use of these medical devices over a longer period of time, the patient receives feedback through the application for medical presentation. This includes the detection of atrial fibrillation recurrences.

SUMMARY:
The present study aims to investigate whether care improvement in patients after catheter ablation/cardioversion compared with standard care can be realized by using a digital eHealth platform with connected mobile sensors through early detection of atrial fibrillation recurrence and patient empowerment.

DETAILED DESCRIPTION:
The main objective of the study is to compare the reliability of detection of atrial fibrillation of 2 measurement methods or protocols in terms of earliest possible detection: (1) digital eHealth platform with tethered 1-lead ECGs vs (2) standard-of-care long-term ECG. In addition, the quality of the acquired ECGs with both protocols will be compared by physician reporting based on the number of false positive abnormal findings as well as possible effects of using different mobile 1-lead ECGs.

Secondary goals are the collection of data on patient adherence (e.g., reliability of performing recommended actions such as measuring ECGs, blood pressure and body weight, and taking medications), on the course of the disease, and on the use of the health care system.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Diagnosis of atrial fibrillation according to ICD-10 I48.0, I48.1, I48.2, or I48.9.
* Catheter ablation or cardioversion no more than 72 hours ago at the time of inclusion.
* Possession and use of a smartphone that allows installation and use of the iATROS app.
* Possession of the physical and mental abilities to use and apply the iATROS app.
* Patients undergoing ablation or cardioversion after a confirmed diagnosis of atrial fibrillation.

Exclusion Criteria:

* < 18 years
* No use of a smartphone
* Lack of the physical and mental abilities necessary to use the iATROS app, or to use so-called "apps" on a smartphone or tablet computer in general
* Absolute contraindications:
* Tumor disease
* immunosuppression
* Dementia in an advanced stage
* Any disease associated with a reduced life expectancy of less than 1 year
* Any disease/condition that restricts participation in the study
* Pregnant or breastfeeding patients
* Participation in another clinical trial
* Addictive diseases
* Stroke in the last 3 months
* Transient ischemic attack (TIA) in the last 3 months

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Superiority of the iATROS platform as compared to the standard of care | 12 months to a maximum of 24 months
  Assessment of atrial fibrillation recurrences and attribution to detection system.
  Clinically relevant superiority of one system over the other is defined at an allocation of ≥75% of all arrhythmic events to either system.

OTHER OUTCOMES:
Patient adherence | 12 months to a maximum of 24 months
  Determination of patient compliance using completion rates of therapy tasks in %
  Collection of data on patient adherence, disease progression, and use of the health care system
Disease progression | 12 months to a maximum of 24 months
  Measurement of blood pressure level progression for hypertensive patients in mmHg
EHRA-Score | Baseline and study completion, an average of 1 year
  Measure of
  - EHRA-Score (European Heart Rhythym Association - Score, possible levels I to IV, with a higher level indicating a higher burden)
Usage of iATROS platform | 12 months to a maximum of 24 months
  Measurement of patient interaction with the provided eHealth solution platform (iATROS platform), with usage being defined as sessions and session length
Health services usage | 12 months to a maximum of 24 months
  Number of
  * patient-doctor interactions
  * ER visits
  * number of in-patient stays for cardiovascular cause
  * number of in-patient stays for non-cardiovascular cause(s)
  * number of out-patient visits for cardiovascular causes at the hospital and/or resident cardiologists
Disease progression | 12 months to a maximum of 24 months
  Number and type of newly diagnosed diseases, with and without cardiovascular cause
Assessment of hsTropI levels | Baseline and study completion, an average of 1 year
  Assessment of heart tissue damage through measure of high sensitive TroponinI (hsTropI) laboratory assay in venous blood in pg/ml
CHA2-DS2-VASc-Score | Baseline and study completion, an average of 1 year
  Measure of
  - CHA2-DS2-VASc-Score (possible levels 0 to 9, with a higher level indicating higher risk)
HASBLED-Score | Baseline and study completion, an average of 1 year
  Measure of
  - HASBLED-Score (possible levels 0 to 9, with a higher level indicating higher risk)
NYHA-classification | Baseline and study completion, an average of 1 year
  Measure of
  - New York Heart Association-classification (possible levels class I to IV, with a higher level indicating higher burden)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Internistisches Zentrum Ebersberg, Ebersberg, Bavaria
  - Isar Herz Zentrum, ISAR Klinikum, Munich, Bavaria
  - Klinikum rechts der Isar of the Technical University of Munich, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: No